## **CONSENT FORM**

## Title of Project: A scalable solution for delivery of Diabetes Self-Management Education in Thailand

Name of PI/Researcher responsible for project: Statement Please initial or thumbprint\* each I confirm that I have read and understood the information sheet. dated 08.10.2018 (version 1.0) for the above named study. I have had the opportunity to consider the information, ask questions and have these answered satisfactorily. I understand that my consent is voluntary and that I am free to withdraw this consent at any time without giving any reason and without my medical care or legal rights being affected. I understand that relevant sections of my/the participant's medical notes and data collected during the study may be looked at by authorised individuals from Chiang Mai University, where it is relevant to my taking part in this research. I give permission for these individuals to have access to these records. I understand that data about/from me/the participant may be shared via a public data repository or by sharing directly with other researchers, and that I will not be identifiable from this information I understand that the tissue sample collected from me will be used to support other research in the future, and may be shared anonymously with other researchers, for their ethically-approved projects I give permission for a copy of this consent form, which contains my personal information, to be made available to the Trial Coordinating Centre for monitoring purposes only. I agree to my health care provider being informed of my participation in the study. agree to me taking part in the above named study. Printed name of participant/Representative Signature of participant/Representative Date (or thumbprint/mark if unable to sign) Printed name of person obtaining consent Signature of person obtaining consent Date The participant is unable to sign. As a witness, I confirm that all the information about the trial was given and the participant/representative consented to taking part (\*only required if the participant/representative is unable to read or write)

Printed name of impartial witness\*

Signature of impartial witness\*

Date